CLINICAL TRIAL: NCT01400542
Title: Sleep Apnea in Early to Mid-Stage Alzheimer's Disease: What Impact of Treatment on the Cognitive Functions of Elderly Patients With Memory Loss?
Brief Title: Sleep Apnea in Early to Mid-Stage Alzheimer's Disease
Acronym: AZAP
Status: Terminated | Type: Observational
Why Stopped: End of the study because of the inclusions were too difficult
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association Lyonnaise de Logistique Posthospitalière (Other)
Responsible Party: Sponsor
Other Study IDs: 1002050; 2010-A01003-36 (Other: AFFSAPS)
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Early Onset Alzheimer Disease; Alzheimer Disease; Obstructive Sleep Apnea Syndromes
Keywords: Early Onset Alzheimer Disease; Alzheimer Disease; Sleep Apnea Syndromes; Obstructive Sleep Apnea Syndromes; Cognitive functions; Continuous Positive Airway Pressure (CPAP) treatment
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea Syndromes; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSAS +: Patient with obstructive sleep apnea syndrome (OSAS)detected at the inclusion visit by a polysomnography
  Interventions: Device: CPAP Treatment
- OSAS -: Patient without obstructive sleep apnea syndrome (OSAS)detected at the inclusion visit by a polysomnography
  Interventions: Device: No treatment

INTERVENTIONS:
Device: CPAP Treatment — Patients with obstructive sleep apnea syndrome will be treated by Continuous Positive Airway Pressure (CPAP) at home during all 4 months all nights.
  Other Names: The CPAP devices used are :; PPC ISLEEP 20 (Breas); PPC S8 AUTOSET SPIRIT II AUTO (Resmed); AUTOSET CS2 (Resmed); REMSTAR AUTO M.SERIES (Respironics); REMSTAR PRO M?SERIES (Respironics); PPC SYSTEM ONE AUTO A FLEX (Respironics); PPC SOMNOSMART 2 (Weinmann)
  Groups: OSAS +
Device: No treatment — no treatment
  Groups: OSAS -

SUMMARY:
Obstructive sleep apnea (OSA) is much more common in the elderly than in the young; the latest studies show prevalence between 45% and 62% in individuals over 60. It is even higher in patients with dementia such as Alzheimer patients.

Several trials in elderly patients showed modified cognitive functions, particularly executive and attentional functions, in patients with respiratory sleep disorder. However the benefit of CPAP (Continuous Positive Airway Pressure) ventilation for Alzheimer patients is still controversial, as there are few studies documenting its effects on dementia patients' cognitive abilities, and clinicians appear reluctant to prescribe this type of treatment.

The investigators must keep in mind that Alzheimer patients suffer significant sleep disorders; advanced- stage patients spend 40% of the night awake and are drowsy a large part of the day. In dementia patients, sleep disorder is a major cause of hospitalization and institutionalization. The prevalence of obstructive sleep apnea (OSA) in this population is estimated at over 50%, and appears to be higher the more advanced the dementia. Trials on obstructive sleep apnea syndromes in Alzheimer patients show significatively improved scores on the apnea-hypopnea index (AHI), as well as satisfactory treatment tolerance. However, any impact on cognitive abilities has yet to be demonstrated.

In addition, cardiovascular pathologies such as arterial hypertension, cardiac arrhythmias, and strokes are strongly correlated to OSA. In light of its consequences on morbidity and mortality, OSA should be considered a public health issue.

In this context, the investigators wish to address the impact of CPAP treatment implementation on the cognitive parameters of patients diagnosed with OSA, particularly on their executive functions. This should provide evidence for mid-term assessment of the benefits of CPAP in caring for elderly patients with dementia.

In light of the prevalence of obstructive sleep pathologies in elderly patients reported in various studies and of the potential impact of CPAP treatment on cognitive abilities, the investigators propose a study to evaluate the impact of OSA treatment on elderly Alzheimer patients' cognitive abilities, particularly on their executive functions.

Executive functions are a rather heterogenous group of high-level cognitive processes which enable individuals to adopt a flexible, context-appropriate behavior. They also include planning abilities, working memory, cognitive control, abstract thought, rule learning, selective attention, motor response selection, etc... Executive functions are mainly associated to the functioning of the brain's frontal lobes, although subcortical structures also play a role. When the executive functions are affected by disease, daily life is significantly impeded as the individual becomes unable to perform complex tasks or regulate his/her behavior. Many tests can help evaluate these functions in dementia patients. A number of "ecological" tests, such as the zoo map test from the Behavioural Assessment of the Dysexecutive Syndrome (BADS) arsenal, are quite relevant for evaluating executive functions.

This project aims to improve the daily life of Alzheimer patients with sleep apnea by improving their executive cognitive functions through CPAP treatment.

According to the Paquid's trial, there are 12,400 Alzheimer patients in the French Loire department. [27] The study population will therefore be recruited in the "La Charité" center of CHU Saint-Etienne. The target population is older individuals (≥ 65) suffering from cognitive disorders similar to Alzheimer's disease.

OSA will be diagnosed based on polysomnography, on an outpatient basis. Apnea patients will receive CPAP treatment for 4 months, which is the minimum duration required to implement and accept treatment, and to measure its impact on patients' neurocognitive abilities.

DETAILED DESCRIPTION:
This study's originality lies in that the target population is elderly and has been diagnosed with both Alzheimer's disease and sleep apnea, and in that it focuses on the impact of treatment on these patient's cognitive abilities, particularly on their executive abilities.We aim to provide practitioners with evidence-based arguments for screening and treating sleep apnea in dementia patients in order to care for these patients, whose treatment options are often scarce.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer-type dementia confirmed by the study's memory specialist.
* MMS comprised between 20 and 28 (inclusive)
* One main caregiver with full mental capacity, living under the same roof, present at all medical visits
* Patient covered by compulsory health insurance
* Patient signed the informed consent form

Exclusion Criteria:

* Prior diagnosis of sleep apnea or patients already benefitting from respiratory assistance equipment- History of COPD (Chronic Obstructive Pulmonary Disease), treated with bronchodilators or corticoids
* Patients with severe heart failure (stages III and IV of the NYHA Functional Classification)
* Patients with a recent history of stroke or myocardial infarction (within the last three months)
* Recently initiated or modified anticholinergic treatment (within the last two months)
* Patients under guardianship
* Behavioral disorders (pacing, agitation)
* Patients with severe dementia
* Patient with potentially low tolerance to treatment (latex allergies, claustrophobia, prior CPAP treatment which was badly tolerated)
* Serious bullous lung disease
* Pneumothorax
* Arterial hypotension
* Dehydration
* Cerebrospinal fluid effusion, recent concussion, or cranial surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with a early or mid-Stage Alzheimer's disease with or without SAOS.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Impact of the CPAP treatment on cognitive functions | At 4 Months
  BADS zoo map scores : subjects are tested in two experimental settings, formulation and execution. The total execution time is the time taken to perform the task assigned in both conditions; the error score measures mistakes made during the test.

SECONDARY OUTCOMES:
Rate of apnea/hypopnea events per hour (AHI/h) | Each month from Day 1 to Month 4
  This secondary outcome measure is only for the treated group by CPAP.
Impact of CPAP treatment on neuropsychological evaluation parameters | At 4 months
  This impact is measured by theses following neuropsychological tests : MMS, clock drawing test, five-word test, Benton Visual Retention Test, Similarities Test (WAIS-R subtest), Coding test (WAIS-III subtest), digit and visual span tasks (forward and backward) from WAIS III, alphabetical and categorical verbal fluency tasks, part A and B of the Trail Making Test, and Stroop test.
  The consideration of these tests separately has no interest. The sum of these tests is important.
Impact of the CPAP treatment on Quality of Life | At 4 months
  It measured by the QOL-AD questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emilie ACHOUR, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No